CLINICAL TRIAL: NCT03597139
Title: An Investigator-Masked, Randomized, Parallel-Group Study of the Ocular Tolerability of Voclosporin Ophthalmic Solution Versus Restasis® in Subjects With Dry Eye Disease
Brief Title: Ocular Tolerability of Voclosporin Ophthalmic Solution Versus Restasis® in Subjects With Dry Eye Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aurinia Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: AUR-VOS-2017-01
Record Dates: First submitted 2018-07-13; First posted 2018-07-24 (Actual); Results first posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-05

CONDITIONS: Dry Eye
Keywords: Dry Eye; Calcineurin Inhibitors
MeSH Terms: conditions — Dry Eye Syndromes | interventions — Cyclosporins

STUDY DESIGN:
Intervention Model Description: This is a Phase 2, multi-center, Investigator-masked, randomized, parallel-group study to evaluate the tolerability, efficacy and safety of VOS versus Restasis® over a 28-day treatment period in subjects with mild to moderate DED. Approximately 90 subjects will be randomized to either VOS or Restasis® at approximately 7 centers located in the US.
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Voclosporin ophthalmic solution (VOS) (Experimental): 0.2% VOS, Twice Daily (BID), both eyes for 28 days
  Interventions: Drug: Voclosporin Ophthalmic Solution
- Comparator (Active Comparator): 0.05% cyclosporine ophthalmic emulsion (Restasis®) BID, both eyes for 28 days
  Interventions: Drug: Restasis®

INTERVENTIONS:
Drug: Voclosporin Ophthalmic Solution — Investigational Drug
  Other Names: 0.2% VOS
  Arms: Voclosporin ophthalmic solution (VOS)
Drug: Restasis® — Comparator
  Other Names: RESTASIS® (cyclosporine ophthalmic emulsion) 0.05%
  Arms: Comparator

SUMMARY:
Evaluate the tolerability, efficacy and safety of VOS versus Restasis® in subjects with mild to moderate Dry Eye Disease (DED).

DETAILED DESCRIPTION:
This is a Phase 2, multi-center, Investigator-masked, randomized, parallel-group study to evaluate the tolerability, efficacy and safety of VOS versus Restasis® over a 28-day treatment period in subjects with mild to moderate DED. Approximately 90 subjects will be randomized to either VOS or Restasis® at approximately 7 centers located in the US

ELIGIBILITY:
Inclusion Criteria:

1. Have a best corrected visual acuity (BCVA) in both eyes of +0.7 logarithm of the Minimum Angle of Resolution (logMAR) or better as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) chart.
2. Have a documented history of DED in both eyes supported by a previous clinical diagnosis.
3. Have ongoing DED, as defined by at least one eye (if one eye, the same eye) meeting all the following criteria:

   * A symptom severity score of ≥30 for Eye Dryness on a Visual Analog Scale (VAS) (0-100)
   * An unanesthetized Schirmer Tear Test (STT) score of ≥1 mm and ≤10 mm per 5 minutes (Note: STT Score obtained at Visit 1)
   * Evidence of ocular surface staining (total fluorescein staining score of at least 3 [0-15 scale]).
4. Have normal lid anatomy.

Exclusion Criteria:

1. Have any known hypersensitivity or contraindication to study treatments (including excipients), topical anesthetics or vital dyes.
2. Be unable to demonstrate correct instillation of over-the-counter (OTC) ocular lubricant.
3. Report discomfort in both eyes from instillation of OTC ocular lubricant during Visit 2 (based on score of ≥30 on the Drop Discomfort VAS).
4. Have used Restasis® (cyclosporine ophthalmic emulsion) within 30 days prior to Visit 1.
5. Have used Restasis® for more than 1 month (if prior use is reported).
6. Have used Xiidra® (lifitegrast ophthalmic solution) within 14 days prior to Visit 1.
7. Have had corneal graft surgery in either eye within 1 year.
8. Have recent or current evidence of ocular infection or inflammation in either eye.
9. Have current evidence of clinically significant blepharitis (defined as requiring lid hygiene therapy), conjunctivitis, or a history of herpes simplex or zoster keratitis in either eye.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2018-08-13 (Actual); Primary Completion 2018-11-09 (Actual); Study Completion 2018-12-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Aurinia Investigative Center, Garden Grove, California
  - Aurinia Investigative Center, Mission Hills, California
  - Aurinia Investigative Center, Rancho Cordova, California
  - Aurinia Investigative Center, Kansas City, Missouri
  - Aurinia Investigative Center, Washington, Missouri
  - Aurinia Investigative Center, High Point, North Carolina
  - Aurinia Investigative Center, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period from August 2018 - December 2018
Period: Overall Study
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Started | 51 | 49
Completed | 47 | 49
Not Completed | 4 | 0
Not completed — Adverse Event | 3 | 0
Not completed — Protocol Non-compliance | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator | Total
Number analyzed (Participants) | 51 | 49 | 100
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (14.51) | 60.2 (15.08) | 58.9 (14.78)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42 | 38 | 80
  Male | 9 | 11 | 20
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 13 | 10 | 23
  Not Hispanic or Latino | 38 | 39 | 77
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 8 | 21
  White | 35 | 36 | 71
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 1 | 1 | 2
Duration of Dry Eye Disease [Median (Inter-Quartile Range); unit: years] — Number of years subject has had Dry Eye Disease
  years | 2.85 [1.62 to 6.13] | 2.67 [1.25 to 6.27] | 2.85 [1.45 to 6.14]

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Drop Discomfort Post Dose Instillation on Day 1
Description: Drop Discomfort was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment 1 minute post-instillation on Day 1. The VAS scale is 0 - 100, where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort".
Time Frame: 1-minute Post Dose 1 installation (Day 1)
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | 7.9 (17.95) | 3.5 (13.30)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.1491, ANCOVA; Mean Difference (Final Values) = 4.6, 95% CI 2-sided [-1.7 to 10.9]

2. Secondary Outcome: Change From Baseline in Drop Discomfort Post Dose Instillation on Day 28
Description: Drop Discomfort was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment 1 minute post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no discomfort" and 100 corresponds to "maximal discomfort".
Time Frame: Day 28
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | 11.8 (20.64) | 6.1 (17.79)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.1187, ANCOVA; Mean Difference (Final Values) = 6.1, 95% CI 2-sided [-1.6 to 13.9]

3. Secondary Outcome: Change From Baseline in Burning/Stinging Post Dose Instillation on Day 28
Description: Burning/Stinging was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no burning/stinging" and 100 corresponds to "worst burning/stinging".
Time Frame: Day 28
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -12.3 (33.22) | -20.1 (25.11)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.2128, ANCOVA; Mean Difference (Final Values) = 6.4, 95% CI 2-sided [-3.7 to 16.5]

4. Secondary Outcome: Change From Baseline in Foreign Body Sensation Post Dose Instillation on Day 28
Description: Foreign Body Sensation was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no foreign body sensation" and 100 corresponds to "worst foreign body sensation".
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -19.7 (35.8) | -20.7 (32.95)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.8408, ANCOVA; Mean Difference (Final Values) = -1.1, 95% CI 2-sided [-11.8 to 9.6]

5. Secondary Outcome: Change From Baseline in Photophobia Post Dose Instillation on Day 28
Description: Photophobia was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no photophobia" and 100 corresponds to "worst photophobia".
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -23.1 (26.35) | -26.2 (25.91)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.5356, ANCOVA; Mean Difference (Final Values) = 2.8, 95% CI 2-sided [-6.1 to 11.6]

6. Secondary Outcome: Change From Baseline in Eye Pain Post Dose Instillation on Day 28
Description: Eye pain was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no eye pain" and 100 corresponds to "worst eye pain".
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -13.9 (31.39) | -19.9 (28.62)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.1787, ANCOVA; Mean Difference (Final Values) = 5.7, 95% CI 2-sided [-2.7 to 14.1]

7. Secondary Outcome: Change From Baseline in Eye Dryness Post Dose Instillation on Day 28
Description: Eye dryness was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no eye dryness" and 100 corresponds to "worst eye dryness".
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -35.0 (27.59) | -34.6 (27.73)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.7666, ANCOVA; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-12.6 to 9.3]

8. Secondary Outcome: Change From Baseline in Itching Post Dose Instillation on Day 28
Description: Itching was assessed using the Individual Symptom Severity Assessment Visual Analog Scale (VAS) where the subject will complete the assessment post-instillation on Day 28. The VAS scale is 0 - 100, where 0 corresponds to "no itching" and 100 corresponds to "worst itching".
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -26.9 (27.41) | -28.1 (30.88)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.8082, ANCOVA; Mean Difference (Final Values) = -1.2, 95% CI 2-sided [-10.7 to 8.4]

9. Secondary Outcome: Change From Baseline in the Total of All Individual Symptom Severity Assessment Scores
Description: The Individual Symptom Severity Assessment Visual Analog Scale (VAS) includes Burning/Stinging (scale 0 - 100; 0 = no Burning/Stinging, 100 = worst Burning/Stinging), Foreign Body Sensation (scale 0 - 100; 0 = no Foreign Body Sensation, 100 = worst Foreign Body Sensation), Photophobia (scale 0 - 100; 0 = no Photophobia, 100 = worst Photophobia), Eye Pain (scale 0 - 100; 0 = no Eye Pain, 100 = worst Eye Pain), Eye Dryness (scale 0 - 100; 0 = no Eye Dryness, 100 = worst Eye Dryness), and Itching (scale 0 - 100; 0 = no Itching, 100 = worst Itching). The total sum of all 6 symptoms (Burning/Stinging, Foreign Body Sensation, Photophobia, Eye Pain, Eye Dryness, Itching) were evaluated (scale 0 - 600; 0 = no visual symptoms, 600 = worst visual symptoms).
Time Frame: Day 28
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm | -130.9 (144.95) | -149.6 (126.16)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Test type: Superiority; p = 0.6362, ANCOVA; Mean Difference (Final Values) = 11.6, 95% CI 2-sided [-37 to 60.3]

10. Secondary Outcome: Change From Baseline in Symptom Assessment in Dry Eye Score (SANDE)
Description: The Symptom Assessment in Dry Eye (SANDE) is a subjective rating performed by the subjects for the frequency and severity of their dry eye symptoms. The total length of the line is 100mm. For Frequency of Symptoms 0mm = "rarely" and 100mm = "all the time". For Severity of Symptoms 0mm = "very mild" and 100mm = "very severe". Subjects were asked to subjectively rate the frequency and severity of their symptoms by placing an "X" on the relevant horizontal line. The length of the line between the "rarely" or "very mild" starting point and the first point where the subject's mark crosses each line was measured and recorded in millimeters.
Time Frame: Day 28
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm
  Frequency | -28.0 (29.37) | -37.9 (27.24)
  Severity | -24.9 (34.06) | -36.1 (24.84)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Frequency; Test type: Superiority; p = 0.0961, ANCOVA — Frequency; Mean Difference (Final Values) = 9.6, 95% CI 2-sided [-1.7 to 20.9]
Statistical Analysis 2: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Severity; Test type: Superiority; p = 0.1722, ANCOVA; Mean Difference (Final Values) = 7.7, 95% CI 2-sided [-3.4 to 18.7]

11. Secondary Outcome: Change From Baseline in Unanesthetized Schirmer Test Score
Description: The Schirmer Test Score recorded tear production on test strips. The Schirmer tear test was conducted 1 hour following administration of VOS/Comparator and 20 minutes following fluorescein corneal staining. Using a ruler and/or the millimeters recorded on the strips, a point halfway between the two lines was measured and this was recorded as the amount of wetting. Lower scores indicate less tear production and therefore a worse outcome. Normal tear production is ≥10mm of wetting on the test strip, and severe dry eye is <5mm of wetting on the test strip.
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm
  Left Eye | 8.5 (10.52) | 3.0 (9.03)
  Right Eye | 8.2 (10.64) | 3.3 (8.39)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Left Eye; Test type: Superiority; p = 0.0051, ANCOVA — Left Eye; Mean Difference (Final Values) = 5.2, 95% CI 2-sided [1.6 to 8.9]
Statistical Analysis 2: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Right Eye; Test type: Superiority; p = 0.0104, ANCOVA — Right Eye; Mean Difference (Final Values) = 4.8, 95% CI 2-sided [1.1 to 8.4]

12. Secondary Outcome: Change From Baseline in Fluorescein Corneal Staining (FCS) Score
Description: The FCS score was summarized for each eye separately. Each of the 5 sections of cornea (superior, inferior, nasal, temporal, central) were graded using the National Eye Institute (NEI) scale; 0, 1 (mild), 2 (moderate), or 3 (severe). The total score was obtained by summing each of the 5 sections of the cornea from 0 - 15. Lower scores indicate less staining and therefore a better outcome.
Time Frame: 28 days
Population: Intent to Treat
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
Number analyzed (Participants) | 51 | 49
mm
  Left Eye | -2.2 (2.90) | -0.2 (3.05)
  Right Eye | -2.2 (3.15) | -0.7 (2.79)
Statistical Analysis 1: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Left Eye; Test type: Superiority; p = 0.0003, ANCOVA — Left Eye; Mean Difference (Final Values) = -2.1, 95% CI 2-sided [-3.2 to -1.0] — Add in RE LE info
Statistical Analysis 2: Comparison: Voclosporin Ophthalmic Solution (VOS) vs Comparator; Right Eye; Test type: Superiority; p = 0.0038, ANCOVA — Right Eye; Mean Difference (Final Values) = -1.6, 95% CI 2-sided [-2.6 to -0.5]

ADVERSE EVENTS:
Time Frame: 28 days +/- 3 days (follow-up period)
Arm/Group | Voclosporin Ophthalmic Solution (VOS) | Comparator
All-Cause Mortality (participants affected / at risk) | 0/51 | 0/49
Serious Adverse Events (participants affected / at risk) | 0/51 | 0/49
Other Adverse Events (participants affected / at risk) | 10/51 | 6/49
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Voclosporin Ophthalmic Solution (VOS) (N=51) | Comparator (N=49)
Ocular Discomfort (Eye disorders) | 7 (9) | 5 (5)
Instillation site pain (General disorders) | 3 (3) | 1 (1)
Lacrimation increased (Eye disorders) | 0 (0) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (4):
  • Study Protocol: aur-vos-2017-01-protocol-v1_Redacted (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03597139/Prot_000.pdf
  • Study Protocol: aur-vos-2017-01-protocol-v2_Redacted (2018-06-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT03597139/Prot_001.pdf
  • Study Protocol: aur-vos-2017-01-protocol-v3_Redacted (2018-07-02): https://cdn.clinicaltrials.gov/large-docs/39/NCT03597139/Prot_002.pdf
  • Statistical Analysis Plan (2018-09-13): https://cdn.clinicaltrials.gov/large-docs/39/NCT03597139/SAP_003.pdf